CLINICAL TRIAL: NCT04226729
Title: Quantitative Assessment of the Vison Using Structural and Functional Indicators and Associations With Brain Function
Brief Title: Associations Between Vision and Brain Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: VISION202201
Record Dates: First submitted 2019-12-30; First posted 2020-01-13 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Healthy; Vision; Disorder, Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy group
- Mild visual impairment group
- Moderate and severe visual impairment group

SUMMARY:
Case-control studies and meta-analysis have reported that several ocular features, especially the thickness of the peripapillary retinal nerve fiber layer and visual acuity, are related to the brain degeneration and cognitive impairment. In our study, we aim to quantitatively assess ocular features using structural and functional indicators and define its associations with brain development and intelligence in children.

ELIGIBILITY:
Inclusion Criteria:

* age from 3 to 12 years old

Exclusion Criteria:

* diagnosed with nervous system disease before

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged 3 to 12 years old. Patients who have been diagnosed with nervous system diseases were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
the visual information processing function | recorded at enrollment
  collected with the electroencephalogram
best corrected visual acuity | recorded at enrollment
  collected with visual acuity chart

SECONDARY OUTCOMES:
refractive status | recorded at enrollment
  the refractive status of both eyes
intraocular pressure | recorded at enrollment
  the intraocular pressure of both eyes
fundus picture | recorded at enrollment
  the fundus pictures of both eyes

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D,Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China